CLINICAL TRIAL: NCT02206204
Title: Single-center, Double-blind, Randomized, Placebo- and Positive-controlled, Parallel-group With Nested Cross-over, Multiple-dose, Up-titration Study of the Effects of Selexipag and Its Metabolite ACT-333679 on Cardiac Repolarization in Healthy Male and Female Subjects
Brief Title: Study of Selexipag and Its Metabolite ACT-333679 on Cardiac Repolarization in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: AC-065-106
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Cardiodynamics; Safety; Tolerability; Pharmacokinetics
Keywords: Selexipag; ACT-333679
MeSH Terms: interventions — selexipag; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): Subjects in Group A receive selexipag on Days 3 to 23 and moxifloxacin-matching placebo on Days 2 and 24. Selexipag administered orally, twice a day, for 21 days according to the following multiple dose up-titration regimen: 400 μg on Days 3-5, 600 μg on Days 6-8, 800 μg on Days 9-11, 1000 μg on Days 12-14, 1200 μg on Days 15-17, 1400 μg on Days 18-20, and 1600 μg on Days 21-23 (only morning dose on Day 23).
  Interventions: Drug: selexipag; Drug: moxifloxacin-matching placebo
- Group B1 (Experimental): Subjects in Group B1 receive 400 mg moxifloxacin, orally on Day 2 and moxifloxacin-matching placebo, orally on Day 24. Subjects receive placebo for selexipag, orally on Days 3 to 23.
  Interventions: Drug: placebo for selexipag; Drug: moxifloxacin; Drug: moxifloxacin-matching placebo
- Group B2 (Experimental): Subjects in Group B2 receive moxifloxacin-matching placebo, orally on Day 2 and 400 mg moxifloxacin, orally on Day 24. Subjects receive placebo for selexipag, orally on Days 3 to 23.
  Interventions: Drug: placebo for selexipag; Drug: moxifloxacin; Drug: moxifloxacin-matching placebo

INTERVENTIONS:
Drug: selexipag
  Arms: Group A
Drug: placebo for selexipag
  Arms: Group B1; Group B2
Drug: moxifloxacin
  Arms: Group B1; Group B2
Drug: moxifloxacin-matching placebo

SUMMARY:
This is a single-center, double-blind, randomized, placebo- and positive-controlled, double-dummy, parallel-group, multiple-dose, up-titration study with a nested cross-over comparison between moxifloxacin and placebo in healthy male and female subjects. The primary objective is to demonstrate that selexipag and its metabolite ACT-333679 do not have an effect on cardiac repolarization exceeding the threshold of regulatory concern, at two orally administered dose levels (800 and 1600 μg twice daily) in healthy male and female subjects. Moxifloxacin is included as a positive control.

ELIGIBILITY:
Inclusion Criteria:

* Signed, dated written informed consent prior to any study procedure.
* Ability to communicate well with the investigator in local language, and to understand and comply with the requirements of the study.
* Women of childbearing potential must have had a negative serum pregnancy test at screening and a negative serum pregnancy test on Day -1. Women of childbearing potential must have consistently and correctly used a reliable method of contraception with a failure rate of < 1% per year, been sexually inactive, or have vasectomized partner.
* Healthy based on medical history and assessments performed at screening and on Day -1.
* Body mass index ≥ 18.5 and ≤ 32 kg/m^2 at screening. Body weight at least 50 kg.
* Negative results from urine drug screen at screening and on Day -1 and negative urine alcohol test on Day -1.
* Willing to refrain from alcohol consumption from at least 48 hours prior to clinic admission to the end of study.
* Systolic blood pressure 90-145 mmHg, diastolic blood pressure 50-90 mmHg, and pulse rate 45-90 beats per minute, at screening and Day -1.
* Hematology, blood chemistry, and urinalysis results not deviating from the normal range to a clinically relevant extent at screening and Day -1.

Exclusion Criteria:

* Known hypersensitivity to selexipag, moxifloxacin, or excipients of the drug formulations used in this study.
* Treatment with selexipag or an investigational drug prior to screening within 30 days or 6 half-lives, whichever was longer.
* History or clinical evidence of any disease and/or the existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism, or excretion of selexipag and moxifloxacin.
* Caffeine consumption of equal to or greater than 800 mg per day at screening.
* History of fainting, collapse, syncope, blackouts, orthostatic hypotension, or vasovagal reactions.
* Chronic or relevant acute infections.
* History of relevant allergy / hypersensitivity.
* History of clinical evidence of psychiatric disease, alcoholism, or drug abuse within the 3-year period prior to screening.
* Smoking within the 3 months prior to screening and inability to refrain from smoking during the study.
* Loss of 500 mL or more of blood within 56 days prior to screening.
* Positive results from the hepatitis serology, except for vaccinated subjects at screening.
* Positive results from human immunodeficiency virus serology at screening.
* Previous treatment with any prescribed or over-the-counter medications, with the exception of contraceptives and hormone replacement therapy, within the 2 weeks prior to first study drug administration or 5 half-lives, whichever longer.
* Excessive physical activities within 1 week prior to administration of study drug.
* Any cardiac condition (including ECG abnormalities) or illness with a potential to increase the cardiac risk of the subject or that may affect QTc analysis.
* QTc > 450 ms or > 470 ms for male or female subjects, respectively, at screening and Day -1.
* Clinically relevant abnormalities on ECG, at screening and Day -1.
* Personal or family history of long QT syndrome or hypokalemia.
* Legal incapacity or limited legal capacity.
* Veins unsuitable for intravenous puncture on either arm.
* Any circumstances or conditions, which, in the opinion of the investigator, may affected the subject's participation in the study or compliance with the protocol.
* Pregnant or nursing women.
* Women who plan to become pregnant within 1 month of the end of study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Baseline adjusted placebo corrected change in corrected QTc interval (time interval from beginning of the Q wave until end of the T wave) (ΔΔQTcI) at various time points | 24 days
  Electrocardiograms (ECGs) will be extracted in replicate at predefined timepoints from replicated 12-lead Holter ECGs. Cardiodynamic endpoints will be assessed at steady-state for 800 μg selexipag on Day 11 and at steady-state for 1600 μg selexipag on Day 23. Based on prospective criteria, QTcI will be the primary method for heart rate (HR) correction.

SECONDARY OUTCOMES:
Baseline adjusted placebo corrected change in heart rate at various time points | 24 days
  Electrocardiograms (ECGs) will be extracted in replicate at predefined timepoints from replicated 12-lead Holter ECGs. Cardiodynamic endpoints will be assessed at steady-state for 800 μg selexipag on Day 11 and at steady-state for 1600 μg selexipag on Day 23.
Baseline adjusted placebo corrected change in RR interval (interval from the peak of one QRS complex to the peak of the next) at various time points | 24 days
  Electrocardiograms (ECGs) will be extracted in replicate at predefined timepoints from replicated 12-lead Holter ECGs. Cardiodynamic endpoints will be assessed at steady-state for 800 μg selexipag on Day 11 and at steady-state for 1600 μg selexipag on Day 23.
Baseline adjusted placebo corrected change in PR interval (time interval from the beginning of the P wave to the beginning of the QRS complex) at various time points | 24 days
  Electrocardiograms (ECGs) will be extracted in replicate at predefined timepoints from replicated 12-lead Holter ECGs. Cardiodynamic endpoints will be assessed at steady-state for 800 μg selexipag on Day 11 and at steady-state for 1600 μg selexipag on Day 23.
Baseline adjusted placebo corrected change in QRS interval (time interval from the beginning of the Q wave to the end of the S wave) at various time points | 24 days
  Electrocardiograms (ECGs) will be extracted in replicate at predefined timepoints from replicated 12-lead Holter ECGs. Cardiodynamic endpoints will be assessed at steady-state for 800 μg selexipag on Day 11 and at steady-state for 1600 μg selexipag on Day 23.
Number of time points at which T-wave morphology changes were observed | 24 days
  Electrocardiograms (ECGs) will be extracted in replicate at predefined timepoints from replicated 12-lead Holter ECGs. Cardiodynamic endpoints will be assessed at steady-state for 800 μg selexipag on Day 11 and at steady-state for 1600 μg selexipag on Day 23.
Maximum plasma concentration (Cmax) for selexipag | 24 days
  Blood will be collected by direct venipuncture or via an intravenous catheter placed in a vein in the arm on Days 11 and 23. Samples will be collected immediately prior to morning dosing and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10 and 12 hours post-dosing. Selexipag concentrations will be quantified in plasma samples by liquid chromatography with tandem mass spectrometry. The measured individual plasma concentrations will be used to directly obtain Cmax
Time to reach maximum plasma concentration (tmax) for selexipag | 24 days
  Blood will be collected by direct venipuncture or via an intravenous catheter placed in a vein in the arm on Days 11 and 23. Samples will be collected immediately prior to morning dosing and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10 and 12 hours post-dosing. Selexipag concentrations will be quantified in plasma samples by liquid chromatography with tandem mass spectrometry. The measured individual plasma concentrations will be used to directly obtain tmax
Area under the plasma concentration-time curve (AUCt) for selexipag | 24 days
  Blood will be collected by direct venipuncture or via an intravenous catheter placed in a vein in the arm on Days 11 and 23. Samples will be collected immediately prior to morning dosing and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10 and 12 hours post-dosing. Selexipag concentrations will be quantified in plasma samples by liquid chromatography with tandem mass spectrometry. AUCt will be calculated according to the linear trapezoidal rule, using the measured concentration-time values above the limit of quantification during one dosing interval.
Trough plasma concentration (Ctrough) for selexipag | 24 days
  Blood will be collected by direct venipuncture or via an intravenous catheter placed in a vein in the arm on Days 11 and 23. Samples will be collected immediately prior to morning dosing and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10 and 12 hours post-dosing. Selexipag concentrations will be quantified in plasma samples by liquid chromatography with tandem mass spectrometry. The measured individual plasma concentrations will be used to directly obtain Ctrough
Maximum plasma concentration (Cmax) for ACT-333679 | 24 days
  Blood will be collected by direct venipuncture or via an intravenous catheter placed in a vein in the arm on Days 11 and 23. Samples will be collected immediately prior to morning dosing and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10 and 12 hours post-dosing. ACT-333679 concentrations will be quantified in plasma samples by liquid chromatography with tandem mass spectrometry. The measured individual plasma concentrations will be used to directly obtain Cmax
Time to reach maximum plasma concentration (tmax) for ACT-333679 | 24 days
  Blood will be collected by direct venipuncture or via an intravenous catheter placed in a vein in the arm on Days 11 and 23. Samples will be collected immediately prior to morning dosing and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10 and 12 hours post-dosing. ACT-333679 concentrations will be quantified in plasma samples by liquid chromatography with tandem mass spectrometry. The measured individual plasma concentrations will be used to directly obtain tmax
Area under the plasma concentration-time curve (AUCt) for ACT-333679 | 24 days
  Blood will be collected by direct venipuncture or via an intravenous catheter placed in a vein in the arm on Days 11 and 23. Samples will be collected immediately prior to morning dosing and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10 and 12 hours post-dosing. ACT-333679 concentrations will be quantified in plasma samples by liquid chromatography with tandem mass spectrometry. AUCt will be calculated according to the linear trapezoidal rule, using the measured concentration-time values above the limit of quantification during one dosing interval.
Trough plasma concentration (Ctrough) for ACT-333679 | 24 days
  Blood will be collected by direct venipuncture or via an intravenous catheter placed in a vein in the arm on Days 11 and 23. Samples will be collected immediately prior to morning dosing and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10 and 12 hours post-dosing. ACT-333679 concentrations will be quantified in plasma samples by liquid chromatography with tandem mass spectrometry. The measured individual plasma concentrations will be used to directly obtain Ctrough
Change in systolic blood pressure from baseline up to end of study | up to 29 days
  Blood pressure and pulse rate will be measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand). Measurements will be recorded from the subject in the supine position after having rested for a 5-minute period.
Change in diastolic blood pressure from baseline up to end of study | up to 29 days
  Blood pressure and pulse rate will be measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand). Measurements will be recorded from the subject in the supine position after having rested for a 5-minute period.
Change in pulse rate from baseline up to end of study | up to 29 days
  Blood pressure and pulse rate will be measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand). Measurements will be recorded from the subject in the supine position after having rested for a 5-minute period.
Change in body weight from baseline up to end of study | up to 29 days
  Body weight will be measured using weighing scales with a precision of at least 0.5 kg.
Number of participants with treatment-related electrocardiogram abnormalities up to the end of study | up to 29 days
  Standard 12-lead electrocardiograms (ECGs) will be recorded at screening, on Day -1, Day 11, Day 23, and at end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Hoch, PhD, Study Director — Actelion
Locations (1):
- Covance Clinical Research Unit, Evansville, Indiana, United States